CLINICAL TRIAL: NCT07405268
Title: The Effect of Levodopa-Benserazide Combination on Periodontal Status in Patients With Parkinson's Disease: A Cross-Sectional Study
Brief Title: Evaluation of the Effects of Levodopa-Benserazide Drug Combination on Periodontal Status in Patients With Parkinson's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özlem SARAÇ ATAGÜN, Assoc Prof Dr., Saglik Bilimleri Universitesi
Other Study IDs: OSATAGUN4
Record Dates: First submitted 2026-02-02; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease (PD); Periodontitis; Periodontal Diseases
Keywords: Levodopa; Benserazide; Salivary Cytokines; Oxidative Stress; Inflammation
MeSH Terms: conditions — Parkinson Disease; Periodontitis; Periodontal Diseases; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Parkinson's - Periodontitis: Patients diagnosed with Parkinson's Disease who also have Periodontitis.
- Parkinson's - Healthy: Patients diagnosed with Parkinson's Disease who are periodontally healthy.
- Control - Periodontitis: Systemically healthy participants (non-Parkinson) who have Periodontitis.
- Control - Healthy: Systemically and periodontally healthy participants.

SUMMARY:
The aim of this study is to evaluate the effects of Levodopa-Benserazide drug combination on periodontal status and salivary cytokine levels in patients with Parkinson's disease. The study includes four groups: Parkinson's patients with periodontitis, periodontally healthy Parkinson's patients, participants without Parkinson's with periodontitis, and periodontally healthy participants without Parkinson's. Clinical periodontal parameters (Plaque Index, Gingival Index, Bleeding on Probing, Pocket Depth, and Clinical Attachment Loss) will be recorded. Unstimulated saliva samples will be collected to analyze the levels of TNF-alpha, RANTES, IL-10, IL-13, Total Oxidant Status (TOS), Total Antioxidant Status (TAS), and Malondialdehyde (MDA).

DETAILED DESCRIPTION:
Background and Rationale: Parkinson's Disease (PD) is a progressive neurodegenerative disorder characterized by the degeneration of dopaminergic neurons in the substantia nigra. Chronic inflammation and oxidative stress are considered significant factors in the progression of PD. Levodopa (L-DOPA), combined with Benserazide, remains the most effective pharmacological treatment for managing PD symptoms. Periodontitis is a chronic inflammatory disease that leads to the destruction of tooth-supporting tissues and is associated with elevated levels of local and systemic inflammatory cytokines such as TNF-alpha, IL-10, IL-13, and RANTES. Recent studies suggest a bidirectional relationship between systemic inflammation and neurodegenerative diseases. This study aims to evaluate the effects of the Levodopa-Benserazide drug combination on periodontal status and salivary inflammatory cytokine levels in patients with Parkinson's Disease.

Study Design and Setting: This cross-sectional, case-control study will be conducted in collaboration with the Department of Periodontology at the University of Health Sciences, Gulhane Faculty of Dentistry, and the Department of Neurology at Hacettepe University Faculty of Medicine.

Participants and Groups: The study will include a total of 136 participants divided into four groups (n=34 per group):

Parkinson's patients with periodontitis

Periodontally healthy Parkinson's patients

Systemically healthy participants with periodontitis (Control)

Systemically and periodontally healthy participants (Control)

Diagnosis of Parkinson's Disease will be confirmed based on the United Kingdom Parkinson's Disease Society Brain Bank Criteria.

Exclusion Criteria: Participants will be excluded if they have active smoking habits, diabetes mellitus, history of antibiotic or anti-inflammatory drug use in the last 3 months, periodontal treatment in the last month, use of probiotics or oral antiseptics in the last month, history of radiotherapy/chemotherapy in the last 6 months, presence of fewer than 16 natural teeth, use of removable partial or complete dentures, or inability to give informed consent due to dementia or other cognitive impairments.

Clinical Evaluations: All participants will undergo a comprehensive periodontal examination. Clinical parameters including Plaque Index (PI) (Silness-Löe), Gingival Index (GI) (Löe-Silness), Bleeding on Probing (BOP), Pocket Depth (PD), and Clinical Attachment Loss (CAL) will be recorded using a Williams periodontal probe. Measurements for PD, CAL, and BOP will be taken at six sites per tooth, while PI and GI will be recorded at four sites per tooth.

Biochemical Analysis: Unstimulated whole saliva samples will be collected from all participants between 09:00 and 10:00 AM to minimize circadian rhythm variations. Participants will be asked to refrain from eating, drinking, or oral hygiene procedures for at least one hour prior to collection. Samples will be stored at -80°C until analysis.

Inflammatory cytokines (TNF-alpha, RANTES, IL-10, IL-13) will be analyzed using Enzyme-Linked Immunosorbent Assay (ELISA).

Oxidative stress markers, including Total Oxidant Status (TOS), Total Antioxidant Status (TAS), and Malondialdehyde (MDA), will be measured using spectrophotometric methods.

Statistical Analysis: Data distribution will be assessed using the Kolmogorov-Smirnov test. Differences between groups will be analyzed using ANOVA (for normally distributed data) or appropriate non-parametric tests. Categorical variables will be compared using the Chi-square test. A p-value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease according to United Kingdom Parkinson's Disease Society Brain Bank Criteria (for study group).
* Systemically healthy individuals (for control group).
* Willingness to participate and sign informed consent.

Exclusion Criteria:

* Active smoking.
* Comprehensive periodontal treatment within the last month.
* Oral, respiratory, or digestive system diseases within the last 3 months.
* Fewer than 16 natural teeth.
* Use of full or removable partial dentures.
* Dementia or inability to provide consent.
* Serious active illnesses or substance abuse.
* Antibiotic treatment within the last 3 months.
* Probiotic use within the last month.
* Radiotherapy/chemotherapy within the last 6 months.
* Use of oral antiseptics within the last month.
* Diabetes mellitus.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from the Department of Neurology at Hacettepe University Faculty of Medicine (Parkinson's patients) and the Department of Periodontology at the University of Health Sciences, Gulhane Faculty of Dentistry (Periodontitis patients and healthy controls).
Sampling Method: Non-Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Salivary Inflammatory Cytokine | Day 1
  TNF-alpha,
Salivary Inflammatory Cytokine | Day 1
  RANTES
Salivary Inflammatory Cytokine | Day 1
  IL-10
Salivary Inflammatory Cytokine | Day 1
  IL-13
Salivary Oxidative Stress Levels | Day 1
  Total Oxidant Status (TOS)
Salivary Oxidative Stress Levels | Day 1
  Total Antioxidant Status (TAS)
Salivary Oxidative Stress Levels | Day 1
  Malondialdehyde (MDA)

SECONDARY OUTCOMES:
Clinical Periodontal Parameters | Day 1
  Assessment of Plaque Index (PI)
Clinical Periodontal Parameters | Day 1
  Bleeding on Probing (BOP)
Clinical Periodontal Parameters | Day 1
  Gingival Index (GI)
Clinical Periodontal Parameters | Day 1
  Pocket Depth (PD)
Clinical Periodontal Parameters | Day 1
  Clinical Attachment Loss (CAL)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wei X, Gibiansky L, Wang Y, Fuh F, Erickson R, O'Byrne S, Tang MT. Pharmacokinetic and Pharmacodynamic Modeling of Serum Etrolizumab and Circulating beta7 Receptor Occupancy in Patients With Ulcerative Colitis. J Clin Pharmacol. 2018 Mar;58(3):386-398. doi: 10.1002/jcph.1031. Epub 2017 Nov 26. PMID 29178491
- [Result] Kononen E, Gursoy M, Gursoy UK. Periodontitis: A Multifaceted Disease of Tooth-Supporting Tissues. J Clin Med. 2019 Jul 31;8(8):1135. doi: 10.3390/jcm8081135. PMID 31370168
- [Result] Ye X, Chen J, Eric Irrgang M, Engel M, Dong A, Glotzer SC, Murray CB. Quasicrystalline nanocrystal superlattice with partial matching rules. Nat Mater. 2017 Feb;16(2):214-219. doi: 10.1038/nmat4759. Epub 2016 Sep 26. PMID 27669053